CLINICAL TRIAL: NCT01180114
Title: SUUBI MAKA ("Hope for Families"): A Family-Based Economic Empowerment Model for Orphaned Children in Uganda
Brief Title: Economic Empowerment Program Suubi-Maka
Acronym: Suubi-Maka
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, PhD, Associate Professor of Social Work, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AAAD2525; R34MH081763-02 (NIH)
Record Dates: First submitted 2010-07-14; First posted 2010-08-11 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Poverty
Keywords: economic empowerment model,; orphaned children and youth,; Uganda,; sub-Saharan Africa

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SUUBI-MAKA (Experimental): Involves creating and broadening asset ownership opportunities and life options for children (ages 12 to 15 years) orphaned due to AIDS in Uganda.
  Interventions: Behavioral: Suubi-Maka ('Hope for Families')
- Usual Care (Other): No intervention for asset ownership, development of future planning skills, enhancement of mental health and reduction of risk taking behaviors for children orphaned due to AIDS in Uganda.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Suubi-Maka ('Hope for Families') — Each child in the SUUBI-MAKA condition receive the usual care plus asset focused services, specifically: a matched Child Development Account (CDA); twelve 1-2 hour training sessions on career planning, setting short-term and long-term career goals, and how to save money; and monthly mentorship program with young adult peers (undergraduate students) on life options and how to avoid risk behaviors. In addition, participants receive a 2:1 match for their deposits into the account. Further, participants and their adult caregivers receive specific training on microenterprise development and specifically on how to start an income-generating project using up to 50% of the matched savings. The intervention is delivered over a period of 24 months.
  Other Names: Children's savings account
  Arms: SUUBI-MAKA
Other: Usual Care — Each child in the control condition receives the usual services for orphaned children (counseling, school lunches, and textbooks).
  Other Names: Usual services
  Arms: Usual Care

SUMMARY:
The overall goal of SUUBI-MAKA is to further develop and preliminarily examine a family economic empowerment intervention that creates economic opportunities (specifically Children Development Accounts) for families in Uganda who are caring for children orphaned due to the AIDS pandemic, and to lay groundwork for a bigger study with practice and policy implications for Sub-Saharan Africa.

DETAILED DESCRIPTION:
The study has two specific aims (1) To conduct formative work in order to understand children and families´ ability and interest in participating in a family-level economic empowerment intervention focused on savings and family income generation, and their response to this family-focused economic empowerment approach alongside additional intervention components, including savings for youth education and adult mentorship. (2) Based on formative data (Aim #1), to adapt the intervention and examine issues related to feasibility and preliminary outcome on a small scale in order to prepare for a larger study.

The intervention, SUUBI-MAKA, uses a novel approach by focusing on economic empowerment of families caring for children orphaned due to AIDS. The intervention has three key components (1) it promotes family-level income generating projects (micro-enterprises) which we believe will enhance economic stability, reduce poverty, and enhance protective family processes for youth orphaned by AIDS. (2) It promotes monetary savings for educational opportunities for AIDS-orphaned children. (3) It provides an adult mentor to children. The intervention will be evaluated via a two-group randomized trial. The two groups are SUUBI-MAKA or Usual care for orphaned children. The participating children will be nested within 20 primary schools that will be randomly assigned such that all children from a particular school receive the same intervention.

ELIGIBILITY:
Inclusion Criteria:

1. An AIDS-orphaned child, defined as a child who has lost one or both parents to AIDS;
2. Enrolled in the last two years of primary school (even though possibly not attending regularly);
3. Between the ages of 11 to 16 years;
4. Living within a family.

Exclusion Criteria:

1. Any youth below 11 years or above 16 years at the time of enrollment in the study;
2. Any youth not enrolled in the final two years of primary school;
3. Any youth who does not self-identify as an AIDS-orphan;
4. Any youth not being raised primarily within a family context at the start of the study.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2008-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Savings and asset-accumulation | 12-month post-intervention
  Formal and informal savings, wealth/assets (e.g. livestock, type of housing), and attitudes toward saving
Educational outcomes | 12-month post-intervention
  School enrollment, School attendance, School grades, Educational plans and aspirations
Sexual risk taking | 12-month post-intervention
  Sexual risk taking behavior (onset of sexual intercourse, unprotected sexual intercourse), Intentions to engage in sexual risk behaviors, HIV knowledge
Savings and asset-accumulation | 24-month post-intervention
  Formal and informal savings, wealth/assets (e.g. livestock, type of housing), and attitudes toward saving
Educational outcomes | 24-month post-intervention
  School enrollment, School attendance, School grades, Educational plans and aspirations
Sexual risk taking | 24-month post-intervention
  Sexual risk taking behavior (onset of sexual intercourse, unprotected sexual intercourse), Intentions to engage in sexual risk behaviors, HIV knowledge

SECONDARY OUTCOMES:
Mental health | 12-month post-intervention
  Self-esteem, depression, hopelessness, helplessness
Social and family support | 12-month post-intervention
  Child-caregiver relationship, family cohesion, family communication, family support
Mental health | 24-month post-intervention
  Self-esteem, depression, hopelessness, and helplessness scales
Social and family support | 24-month post-intervention
  Child-caregiver relationship, family cohesion, family communication, family support

CONTACTS AND LOCATIONS:
Overall Officials: Fred M Ssewamala, PhD, Principal Investigator — Columbia University
Locations (1):
- St. Joseph's Matale Parish, Rakai, Rakai, Uganda

REFERENCES:
- [Derived] Tutlam NT, Filiatreau LM, Byansi W, Brathwaite R, Nabunya P, Sensoy Bahar O, Namuwonge F, Ssewamala FM. The Impact of Family Economic Empowerment Intervention on Psychological Difficulties and Prosocial Behavior Among AIDS-Orphaned Children in Southern Uganda. J Adolesc Health. 2023 May;72(5S):S51-S58. doi: 10.1016/j.jadohealth.2023.01.002. PMID 37062584
- [Derived] Jennings L, Ssewamala FM, Nabunya P. Effect of savings-led economic empowerment on HIV preventive practices among orphaned adolescents in rural Uganda: results from the Suubi-Maka randomized experiment. AIDS Care. 2016;28(3):273-82. doi: 10.1080/09540121.2015.1109585. Epub 2015 Nov 7. PMID 26548549
- [Derived] Han CK, Ssewamala FM, Wang JS. Family economic empowerment and mental health among AIDS-affected children living in AIDS-impacted communities: evidence from a randomised evaluation in southwestern Uganda. J Epidemiol Community Health. 2013 Mar;67(3):225-30. doi: 10.1136/jech-2012-201601. PMID 23410851